CLINICAL TRIAL: NCT04851522
Title: The Impact of Dilute Bleach Compresses on the Incidence and Severity of Radiation Dermatitis
Brief Title: Dilute Bleach Compresses for Radiation Dermatitis
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of patient accrual in the past year.
Sponsor: Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Jennifer Huang, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-078
Record Dates: First submitted 2021-04-16; First posted 2021-04-20 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Radiation Dermatitis
Keywords: Radiation Dermatitis
MeSH Terms: conditions — Radiodermatitis | interventions — Sodium Hypochlorite; Petrolatum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Di-Dak-Sol + White Petrolatum (Experimental): Participants will receive Di-Dak-Sol (dilute bleach compresses) prior to receiving radiation. This will continue throughout their radiation therapy and for one week after.
  Participants will also be asked to apply white petrolatum ointment 2x daily throughout treatment: once after radiation and once in the evening.
  Participants will be provided with a log and asked to document information (dates/times of application) about the study treatment .
  Interventions: Drug: Di-Dak-Sol; Other: White Petrolatum

INTERVENTIONS:
Drug: Di-Dak-Sol — Topical solution applied externally.
  Other Names: Sodium Hypochlorite; Diluted NaOCl
Other: White Petrolatum — Topical ointment applied externally
  Other Names: Petroleum jelly; Soft paraffin; Multi-hydrocarbon

SUMMARY:
This study is looking at the safety of applying dilute bleach compresses to patients receiving radiation therapy and the impact of these dilute bleach compresses on the frequency and severity of skin changes that occur during radiation therapy.

The names of the study interventions involved in this study are:

* Di-Dak-Sol: dilute bleach compresses
* White petrolatum ointment

DETAILED DESCRIPTION:
This is a planned open-label prospective clinical trial to determine the safety of applying dilute bleach compresses to pediatric patients being treated for rhabdomyosarcoma and other soft tissue and bone sarcomas with radiation therapy (RT).

This study is interested in finding out whether dilute bleach compresses are safe to apply and evaluating their impact on the frequency and severity of skin changes that occur in children who are receiving radiation therapy for cancer treatment.

This information may help treat other patients receiving radiation therapy for cancer treatment in the future.

The research study procedures include screening for eligibility and study treatment including weekly evaluations and follow up visits

Participants will receive study treatment throughout their radiation therapy and for one week after. They will be followed for one month after the completion of radiation.

It is expected that about 12 people will take part in this research study.

.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with a rhabdomyosarcoma or other sarcoma requiring RT
* 12 to 25 years of age
* Scheduled for a RT planning session (CT simulation)
* Have a scheduled RT start date within 1 to 2 weeks from the CT simulation
* Will be receiving doses of radiotherapy greater than at least 36 Gy
* Subjects may participate in other studies, including therapeutic trials.
* Ability to comply with at-home dilute Di-Dak-Sol compresses for final week of dilute Di-Dak-Sol compresses following radiation treatment.
* Ability to understand and/or the willingness of their parent or legally authorized representative to sign a written informed consent document.

Exclusion Criteria:

* Patients who are pregnant, which may result in discontinuation of RT
* Presence of inflammatory skin lesions in the radiation field that could interfere with assessment

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2021-06-09 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE Version 5.0 | 1 year
  The number and proportion of adverse events, graded as defined by CTCAE version 5.0 will be tabulated by type and grade.

SECONDARY OUTCOMES:
Number of Participants with Radiation dermatitis | 1 year
  Incidence and severity of radiation dermatitis according to CTCAE v5.0 grade analyzed using descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Huang, MD, Principal Investigator — Boston Children's Hospital

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Technology & Innovation Development Office at www.childrensinnovations.org or email TIDO@childrens.harvard.edu Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu